CLINICAL TRIAL: NCT01616485
Title: A Double-blind, Randomized, Crossover Evaluation of the Hemodynamic Response to Sublingual Glyceryl Trinitrate in Patients Receiving TA-1790, Sildenafil, and Placebo
Brief Title: Study to Evaluate Hemodynamic Response to to a Sublingual Dose of Glyceryl Trinitrate in Subjects Receiving TA-1790, Sildenafil Citrate, and Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TA-04
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate; Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment A (Experimental): TA-1790 + glyceryl trinitrate
  Interventions: Drug: TA-1790; Drug: Nitrostat
- Treatment B (Active Comparator): sildenafil citrate + glyceryl trinitrate
  Interventions: Drug: Sildenafil citrate; Drug: Nitrostat
- Treatment C (Placebo Comparator): placebo + glyceryl trinitrate
  Interventions: Drug: Placebo; Drug: Nitrostat

INTERVENTIONS:
Drug: TA-1790 — 2 TA-1790 100 mg capsules
  Arms: Treatment A
Drug: Sildenafil citrate — 2 sildenafil citrate 50 mg capsules
  Arms: Treatment B
Drug: Placebo — 2 placebo capsules for TA-1790 100 mg capsules
  Arms: Treatment C
Drug: Nitrostat — glyceryl trinitrate tablet, USP 0.4 mg

SUMMARY:
The objective of this study is to evaluate the hemodynamic response to a sublingual dose of glyceryl trinitrate in subjects receiving oral TA-1790, sildenafil citrate, and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Willing to comply with all study requirements and clinic schedules
* Male between 30 to 60 years of age
* Non-smoker
* No history of alcohol abuse
* Normal screening laboratory values

Exclusion Criteria:

* Allergy or hypersensitive to PDE5 inhibitors
* Evidence of clinically significant disease
* Supine systolic/diastolic blood pressure level
* History of cardiovascular disease
* Previously participated in TA-1790 within the past 30 days

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2004-03; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Change in hemodynamic measurements | Pre-dose, 5 min interval for first 45 minutes. 60, 90, and 120 minutes post-dose.
  Change in hemodynamic measurements consisted of blood pressure and pulse rate measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Peterson, MS, Study Director — VIVUS LLC
Locations (1):
- MDS Pharma Services, Phoenix, Arizona, United States